CLINICAL TRIAL: NCT05970835
Title: Validation of a Mobile App as an Adjuvant Treatment for Thermal Context Patients: a Randomized Controlled Trial Protocol
Brief Title: Validation of a Mobile App as an Adjuvant Treatment
Acronym: VMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ISAVE- Instituto Superior de Saúde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISAVE
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Validation
Keywords: thermalism; tourism; assessment; clinical
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This will be a single-blinded, parallel two-arm group randomised, controlled, superiority trial with a 3 months of intervention period in real thermal treatment conditions, in Caldelas- Amares, Portugal. The target population will be recruited among the patients who use the thermal environment in Caldelas- Amares.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors and data analysts will remain blinded to participant´s allocation group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Firstly, all patients will be evaluated using Physical Performance Test, Saint George's Respiratory Questionnaire , and Geriatric Pain Measure and the MiniMental Satet Exam to fulfill the eligibility criteria. After that participants will be randomly assigned using the software www.randomizer.org. to control or intervention group. Outcome assessors and data analysts will remain blinded to participant´s allocation group.
  Participants assigned to control group will receive the usual care provided by clinicians and physiotherapists from the Complexo Termal de Caldelas. They will have an educational session conducted by one of the researchers, and a paper sheet will be distributed with exercises and a written explanation of how to perform those exercises and the number of sets and repetitions.
  Interventions: Other: Control group
- Experimental group (Experimental): Concerning patients from the intervention group will have an educational session given by one of the researchers, explaining how to use the HealthSmArt_ISAVE App. Then each patient will be given a unique code and password to log into the App and to start working with their smartphones. HealthSmArt_ISAVE App has three main components which are: evaluation (short, medium and long term); screening and intervention/rehabilitation.
  Interventions: Other: Experimental group

INTERVENTIONS:
Other: Control group — Participants assigned to control group will receive the usual care provided by clinicians and physiotherapists from the Complexo Termal de Caldelas. Participants will have an educational session conducted by one of the researchers, and a paper sheet will be distributed with exercises and a written explanation of how to perform those exercises and the number of sets and repetitions. data collection will be conducted in moments t2 and t3 by a phone call.
  Arms: Control group
Other: Experimental group — Experimental group evaluation: balance, functionality- 30 Second Sit To Stand Test, Modified Medical Research Council and functional status questionnaire, pain using VAS, cognitive variables-Montreal Cognitive Assessment and self-reported thermal water effects.After evaluation the App will display exercises related to data collected. Outcome measures will be collected at baseline, and 1 week, 1 month and 3 months after baseline.
  After evaluation the App will display exercises related to data collected concerning participants condition improvement.
  Arms: Experimental group

SUMMARY:
Health tourism is one of the most important touristic activities. It can generate economic and social value. Balneotherapy is one of the options concerning healthcare and well-being. Although this fact it lacks information concerning effectiveness of thermal water treatments. Digital Technologies are being implemented and developed in health care systems, stimulated also by World Health Organization (WHO), in order to facilitate and improve patients' treatment and assessment. Traditional approach does not allow a follow-up due to the fact the patient leaves the thermal complex after treatment or several other reasons due to that the gap persists and social security of each country avoids support based on this lack of information. It is important to fulfil this gap and for that digital technologies seem to be the answer.

This study aims to investigate effectiveness in self-management and clinical assessment and monitorization between a smartphone app (HealthSmArt_ISAVE) and a standard approach.

DETAILED DESCRIPTION:
This will be a single-blinded, parallel two-arm group randomised, controlled, superiority trial with a 12 months of intervention period in real thermal treatment conditions, in Caldelas, Amares, Portugal. The target population will be recruited among the patients who use the thermal environment in Caldelas- Amares.

The random sequence, with a 1:1 allocation of participants in control and intervention groups is going to be generated using an external website. The outcome data will be collected from stored data by a research assistant who is blinded to the treatment arm.

The study will be supported by clinicians, physiotherapists, and psychologists and will be developed in ISAVE in partnership with Complexo Termal de Caldelas.

The guideline SPIRIT (Standard Protocol Items: Recommendations for Interventional Trials) will be used for report elaboration and the manuscript will follow CONSORT (Consolidated Standards for Reporting Trials) guidelines for the transparent reporting of randomized trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults, in treatment at Complexo Termal de Caldelas- Amares, Portugal,
* with chronic musculoskeletal problems
* respiratory issues
* with satisfactory cognitive analysis for exercise

Exclusion Criteria:

* having received intramuscular or intraarticular steroid injections within 4 weeks, pregnancy, moderate or severe cognitive impairment

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Balance evaluation | From baseline until the last up to 9 months
  Balance will be evaluated using Berg Balance Scale, composed by 14 items, Item-level scores range from 0-4, determined by ability to perform the assessed activity, Item scores are then summed, Maximum score = 56
Functional ability | From baseline until the last up to 9 months
  The participant is encouraged to complete as many full stands as possible within 30 seconds.

SECONDARY OUTCOMES:
Dyspnea | Through the study completion, an average 1 year
  evaluation of dyspnea using Modified Medical Research Council (mMRC) breathlessness scale ranges from grade 0 to 4.
Evaluate pain | through study completion, an average of 1 year
  evaluation of pain and morning stiffness, using visual analog scale, considering 1 the lowest pain ever felt and 10 the worst pain ever felt

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ribeiro, PhD, Principal Investigator — ISAVE- CICS
Locations (1):
- ISAVE, Amares, Braga District, Portugal

IPD SHARING:
Plan to Share IPD: No